CLINICAL TRIAL: NCT04037293
Title: Premature Atherosclerosis in Systemic Lupus Erythematosus: a Prospective Cohort Study
Brief Title: Premature Atherosclerosis in Systemic Lupus Erythematosus
Acronym: PASLE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: JS-2057
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: SLE; Atherosclerosis
Keywords: SLE; Atherosclerosis; carotid intima media thickness; brachial-ankle pulse wave velocity; risk factors; Cohort
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — 1.5ml blood plasma will be retained from each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CIMT and baPWV measurement — All patients will receive carotid intima media thickness (CIMT) and brachial-ankle pulse wave velocity (baPWV) measurement at baseline and 5-year follow-up.

SUMMARY:
Patients with SLE have increased rates of atherosclerosis, while the risk factors for atherosclerosis in those patients were not fully revealed. This study is an observational study to investigate the natural process and risk factors for atherosclerosis based on a Chinese SLE cohort. Carotid intima media thickness (CIMT) and brachial-ankle pulse wave velocity (baPWV) will be measured for each patient at baseline and 5-year follow-up. Blood tests including cholesterol levels, fasting plasma glucose levels and etc. will also be performed.

DETAILED DESCRIPTION:
Accelerated atherosclerosis is a major complication of systemic lupus erythematosus (SLE), and it leads to increased cardiovascular morbidity and mortality in patients with SLE. Prevention and intervention of premature atherosclerosis is beneficial for prognosis and survival of patients with SLE.

The primary aim of this study was to investigate the natural progress of carotid intima media thickness (CIMT) in 5 years, and examine the risk factors for progression of CIMT and atherosclerotic plaques based on a Chinese SLE cohort. The secondary aims of the study were to investigate progression of brachial-ankle pulse wave velocity (baPWV), and to examine the risk factors for increasing baPWV in patients with SLE.

Based on sample size calculation, 440 patients who meet the eligibility criteria will be enrolled in this study. All patients will be enrolled from Peking Union Medical College Hospital. After informed consent is obtained, the patients will be comprehensively evaluated from demographic characteristics, medical history, clinical assessments, laboratory tests results, CIMT and baPWV at baseline and 5-year follow-up. Descriptive analysis, univariate analysis, and multivariate analysis will be used to analyze the correlation between potential risk factors and CIMT/baPWV.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Fulfillment of clinical classification criteria of SLE (four or more 1997 American College of Rheumatology classification criteria)
* Provision of signed written informed consent

Exclusion Criteria:

* Clinically overt coronary artery disease
* A history of cardiovascular disease (previous stroke, heart failure, myocardial infarction, angina, or symptomatic PAD)
* Malignancy
* Pregnant/lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population was patients with the clinical diagnosis of SLE. Study participants were recruited through a nationwide registry system created by the Chinese SLE Treatment and Research group. All patients were continuously enrolled as outpatients of the Department of Rheumatology in Peking Union Medical College Hospital (PUMCH), which is a renowned hospital in China.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
quantitative change in CIMT from baseline | Year 5
  quantitative changes in CIMT at 5-year follow-up from baseline will be documented

SECONDARY OUTCOMES:
quantitative change in baPWV from baseline | Year 5
  quantitative changes in baPWV at 5-year follow-up from baseline will be documented
Major cardiovascular events | 5 years
  the prevalence rate of nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Shuyang Zhang, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hostipal, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giannelou M, Mavragani CP. Cardiovascular disease in systemic lupus erythematosus: A comprehensive update. J Autoimmun. 2017 Aug;82:1-12. doi: 10.1016/j.jaut.2017.05.008. Epub 2017 Jun 9. PMID 28606749
- [Background] Esdaile JM, Abrahamowicz M, Grodzicky T, Li Y, Panaritis C, du Berger R, Cote R, Grover SA, Fortin PR, Clarke AE, Senecal JL. Traditional Framingham risk factors fail to fully account for accelerated atherosclerosis in systemic lupus erythematosus. Arthritis Rheum. 2001 Oct;44(10):2331-7. doi: 10.1002/1529-0131(200110)44:103.0.co;2-i. PMID 11665973
- [Background] Manzi S, Meilahn EN, Rairie JE, Conte CG, Medsger TA Jr, Jansen-McWilliams L, D'Agostino RB, Kuller LH. Age-specific incidence rates of myocardial infarction and angina in women with systemic lupus erythematosus: comparison with the Framingham Study. Am J Epidemiol. 1997 Mar 1;145(5):408-15. doi: 10.1093/oxfordjournals.aje.a009122. PMID 9048514